CLINICAL TRIAL: NCT02503007
Title: The Effects of 14-days of HMB-Free Acid on Changes in Muscle Architecture, Blood Markers of Muscle Damage and Performance During 4-Days of Survival Training
Brief Title: Effects of 14-days of HMB-free Acid on Changes in Muscle During 4-days of Survival Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Koach Sport and Nutrition (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: MTI2015-CS01
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Survival Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): A placebo similar in composition and appearance to the experimental treatment.
  Interventions: Dietary Supplement: Placebo
- HMB-FA (Experimental): Active treatment consisting of 3 g of HMB-FA per day.
  Interventions: Dietary Supplement: HMB-FA

INTERVENTIONS:
Dietary Supplement: Placebo
  Arms: Placebo
Dietary Supplement: HMB-FA
  Other Names: beta-hydroxy-beta-methylbutyric acid
  Arms: HMB-FA

SUMMARY:
Sustained high-intensity activity, such as survival training with little nourishment available, can result in a loss of muscle performance. This study will examine the effects of a nutritional supplement to maintain muscle and muscle performance during this period.

DETAILED DESCRIPTION:
Sustained high intensity activity that is often accompanied by sleep and nutrient deprivation is a common characteristic of survival training. Survival training is a requirement in the preparation of pilots, where they learn evasion and survival skills that they may need to avoid capture in a situation in which they have bailed from their plane. The physiological stresses associated with the nature of these operations often results in significant decrements in lean body mass, muscle size and muscle endurance and power. During a sudden evacuation from the aircraft the pilot only takes a small survival bag. There is a limit to what can possibly be put in this bag. However, the ability to provide a dietary supplement specifically targeting muscle may provide an important resource for maintaining muscle mass and performance. Thus, the purpose of this study is to determine the efficacy of 14 days of HMB-FA ingestion on maintaining muscle architecture and muscle performance during 4-days of survival training. In addition, anabolic and catabolic markers of stress, inflammation and muscle damage will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 27 Years of age
* Soldier members of Special Operations
* Healthy as assessed by the Unit's Medical Officers
* Subject provides written and dated informed consent to participate

Exclusion Criteria:

* A history of medical or surgical events that may significantly affect the study outcome, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders
* Use of medications that may affect the study outcomes
* Use of nutritional supplements (such as protein drinks, creatine, HMB and vitamins) in the 3 months prior to the start of the study
* Subject is currently participating in another clinical trial or has received an investigational product within thirty days prior to screening/enrollment

Ages: 18 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Day 18
  Hand grip strength will be measured using a hand-grip dynamometer.

SECONDARY OUTCOMES:
Muscle Power | Day 18
  Vertical Jump power will be measured using a linear transducer.
Muscle Morphology | Day 18
  Muscle morphology will be measured using a 3.0 Tesla Magnetic Resonance Imaging device.
Muscle Mass | Day 18
  Muscle mass will be performed using bioelectrical impedance
Blood Biochemical Analysis | Day 18
  Blood biochemical analysis will be performed using an ELISA assay.
Urine Biochemical Analysis | Day 18
  Urine biochemical analysis will be performed using an ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Ishay Osterfeld, MD, Principal Investigator — International Diabetes Federation
Locations (1):
- IDF, Beersheva, Israel